CLINICAL TRIAL: NCT03241160
Title: The Severity of Chewing Disorders is Related to Gross Motor Function and Trunk Control in Cerebral Palsy
Brief Title: Chewing Disorders, Gross Motor Function and Trunk Control in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Other Study IDs: HACETTEPE
Record Dates: First submitted 2017-08-02; First posted 2017-08-07 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cerebral palsy: Children with a diagnosis of spastic cerebral palsy aged between 2 to 12 years who will be referred by pediatric neurologists will be included. Children under the age of 24 months, and used any medicine and/or oral appliances that could affect the chewing performance, will be excluded. Chewing evaluation will be performed.
  Interventions: Other: Chewing evaluation

INTERVENTIONS:
Other: Chewing evaluation — Chewing evaluation will be performed. An experienced physical therapist who will take a scale training session will do the chewing evaluation according to the chewing performance scale.This scale classifies chewing function on an ordinal scale with five levels between 0 and 4 based on the sequence of functional movements during chewing.

SUMMARY:
The study is planned to determine the relationship between chewing performance level and gross motor function, and trunk postural control in cerebral palsy (CP).

DETAILED DESCRIPTION:
The study is planned to determine the relationship between chewing performance level and gross motor function, and trunk postural control in cerebral palsy (CP). Chewing performance level will be determined by the chewing performance scale. The Gross Motor Function Classification System (GMFCS) will be used to determine gross motor function levels. Segmental Assessment of Trunk Control (SATCo) will be used to measure trunk control. The correlations between chewing performance level and gross motor function, and trunk postural control will be assessed. The Chi-square test will also be used to compare GMFCS levels and trunk control in children with and without chewing disorders.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of cerebral palsy
* Referring by a pediatric neurologist
* Aging between 2 to 12 years

Exclusion Criteria:

* Aging under the age of 24 months
* Using any medicine and/or oral appliances that could affect the chewing performance

Ages: 2 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Children with a diagnosis of spastic cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2017-09-08 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Chewing evaluation | 15 days
  Chewing evaluation will be determined by a scale that classifies chewing function on an ordinal scale with five levels between 0 and 4 based on the sequence of functional movements during chewing.

SECONDARY OUTCOMES:
Gross motor function evaluation | 15 days
  Gross motor function evaluation will be performed according to the Gross Motor Function Classification System.
Trunk control evaluation | 15 days
  Segmental Assessment of Trunk Control (SATCo) will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serel Arslan S, Demir N, Inal O, Karaduman AA. The severity of chewing disorders is related to gross motor function and trunk control in children with cerebral palsy. Somatosens Mot Res. 2018 Sep-Dec;35(3-4):178-182. doi: 10.1080/08990220.2018.1521788. Epub 2018 Dec 28. PMID 30592431